CLINICAL TRIAL: NCT00337974
Title: Computer-Based Training for Cognitive Enhancement: In Home Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OUT-106-2005
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Aging
Keywords: cognitive enhancement; memory; auditory memory; speech; computerized
MeSH Terms: conditions — Speech

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental Treatment (Experimental): Computerized Plasticity-Based Adaptive Cognitive Training
  Interventions: Other: Computerized Plasticity-Based Adaptive Cognitive Training
- Active Control (Active Comparator): Educational DVDs
  Interventions: Other: Educational DVDs
- No Contact Control (No Intervention)

INTERVENTIONS:
Other: Computerized Plasticity-Based Adaptive Cognitive Training
  Other Names: BrainHQ; Brain Fitness Program
  Arms: Experimental Treatment
Other: Educational DVDs
  Arms: Active Control

SUMMARY:
The primary objective of this study is to evaluate the effects of a computer-based training program on the memory and cognitive abilities of mature individuals undergoing healthy aging.

DETAILED DESCRIPTION:
The computer-based training program is focused on speech reception to strengthen an individual's memory for speech. This type of training program was chosen because speech perception and memory are crucial elements of human communication and losses in this area are often the first signal of overall cognitive decline.

Subjects meeting eligibility criteria and providing written, informed consent are randomized to three groups; two 40-session, computerized training programs or a no contact control group.

ELIGIBILITY:
Inclusion Criteria:

A)Participants must be at least 60 years old B)Participants must have a Mini-Mental State Exam (MMSE) score of 24 or higher to ensure that participants do not meet common criteria for dementia C)Participants must be a native English speaker D)Participants must be able to see well enough to read the consent form E)Participants must be able to hear well enough to understand ordinary spoken conversation in a slightly noisy room F)Participants must be willing to commit to the time requirements of the study and not have any scheduled trips or absences for more than 1 week during the training.

Exclusion Criteria A)Participants must not be planning to begin cholinesterase inhibitor (AChEI) therapy or to change their dosing levels. Subjects currently using AChEI will be included if they have an established steady dosing history at least one month prior to the study and are expected to continue at the same dosage throughout the study.

B)Participants must not have had a head trauma that caused them to lose consciousness.

C)Participants must not have had a stroke within the past year; or have had a stroke that has left them with expressive or receptive language problems.

D)Participants must not have any central nervous system disorder that could contribute to cognitive impairment.

E)Participants must not have a tremor preventing the use of a computer mouse or other pointing device.

F)Participants must not currently be active in another clinical trial.

Exclusion Criteria:

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2005-03; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of training effects.

SECONDARY OUTCOMES:
Safety effects of computer-based training.

CONTACTS AND LOCATIONS:
Overall Officials: Henry W Mahncke, PhD, Principal Investigator — Posit Science Corporation
Locations (1):
- Posit Science Corporation, San Francisco, California, United States

REFERENCES:
- [Result] Mahncke HW, Connor BB, Appelman J, Ahsanuddin ON, Hardy JL, Wood RA, Joyce NM, Boniske T, Atkins SM, Merzenich MM. Memory enhancement in healthy older adults using a brain plasticity-based training program: a randomized, controlled study. Proc Natl Acad Sci U S A. 2006 Aug 15;103(33):12523-8. doi: 10.1073/pnas.0605194103. Epub 2006 Aug 3. PMID 16888038